CLINICAL TRIAL: NCT04340856
Title: Retrospective, Uncontrolled Multcentric Cohort Study on the Therapy of Chronic Megalon (CoMeC)
Brief Title: Retrospective, Uncontrolled Cohort Study on the Therapy of Chronic Megalon
Acronym: CoMeC
Status: Completed | Type: Observational
Sponsor: Theresienkrankenhaus und St. Hedwig-Klinik GmbH (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: Chronic Megacolon 001
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Megacolon
Keywords: Megacolon
MeSH Terms: conditions — Megacolon | interventions — Colectomy; Laxatives; polyethylene glycol 3350; Bisacodyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: colon surgery — There are no guidelines to direct surgical therapy in patients with chronic megacolon. Historically, it is the surgeons individual choice to use one of the above mentioned surgical treatments. Therefore, the aim of this study is to analyze the success and downsides of the different surgical approaches.
  Other Names: Subtotal colectomy with ileorectal anastomosis; Diverting loop ileostomy; Colectomy with ileoanal anastomosis; Decompressive cecostomy with periodic antegrade enemas; Segmental colon resection
Drug: Laxatives — There are no guidelines to direct laxative measures in patients with chronic megacolon. Historically, it is the gastroenterologists individual choice to use one of the above mentioned laxative measures. Therefore, the aim of this study is to analyze the success and downsides of the different Laxative measures.
  Other Names: High-colonic water enema; Water-soluble contrast enema; PEG electrolyte solution; Colon decompression probe; Prucaloprid; Bisacodyl

SUMMARY:
The aim of this retrospective cohort study is to analyze all available data of patients with chronic megacolon in three clinical centers with respect of conservative and surgical therapies.

DETAILED DESCRIPTION:
Megacolon may be defined as dilatation of the abdominal colon with a minimum of 9 cm in diameter and the absence of mechanical obstruction. Chronic megacolon in adults is an acquired uncommon condition that generally is associated with constipation. It has to be distinguished from other forms of megacolon such as acute toxic megacolon, acute non-toxic megacolon (Ogilvie´s-syndrome) and congenital megacolon (Hirschsprung disease). Regardless of concomitant diseases and causes, most patients with chronic megacolon were treated by laxative measures. Less is known about the optimal conservative therapy . If conservative measures fail, there are several surgical options, depending upon anorectal function. However, less in known about the optimal surgical therapy of patients with chronic megacolon. The aim of this retrospective cohort study is to analyze all available data of patients with chronic megacolon in three clinical centers with respect of conservative and surgical therapies.

ELIGIBILITY:
Inclusion Criteria:

* Chronic megacolon (colon diameter > 90 mm)

Exclusion Criteria:

* Toxic megacolon
* Ogilvie-syndrome
* Hirschsprung disease
* Mechanical colorectal obstruction

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The databases of three clinical centers were systematically screened for patients with chronic megacolon (exclusion/inclusion criteria) in the time frame from 1.5.2005 to 1.5.2020.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Constipation | One year after inpatient treatment (conservative/surgery)
  Number of constipation crises leading to further hospital admissions: n

SECONDARY OUTCOMES:
Hospital stay | Three months after inpatient treatment (conservative/surgery)
  Hospital stay after inpatient treatment (conservative/surgery): days
Adverse events | 30 days after inpatient treatment (conservative/surgery)
  Any adverse event after inpatient treatment (conservative/surgery): n

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Schmitz, PhD, MD, Principal Investigator — Theresienkrankenhaus und St.Hedwigkliniken Mannheim,University of Heidelberg
Locations (1):
- Theresienkrankenhaus und St. Hedwigkliniken GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanauer SB, Wald A. Acute and chronic megacolon. Curr Treat Options Gastroenterol. 2007 Jun;10(3):237-47. doi: 10.1007/s11938-007-0017-z. PMID 17547862
- [Background] O'Dwyer RH, Acosta A, Camilleri M, Burton D, Busciglio I, Bharucha AE. Clinical Features and Colonic Motor Disturbances in Chronic Megacolon in Adults. Dig Dis Sci. 2015 Aug;60(8):2398-407. doi: 10.1007/s10620-015-3645-5. Epub 2015 Apr 14. PMID 25868630
- [Background] Wang XJ, Camilleri M. Chronic Megacolon Presenting in Adolescents or Adults: Clinical Manifestations, Diagnosis, and Genetic Associations. Dig Dis Sci. 2019 Oct;64(10):2750-2756. doi: 10.1007/s10620-019-05605-7. Epub 2019 Apr 5. PMID 30953226
- [Derived] Schmitz D, Meier E, Axt S, Arlt G, Kienle P, Johannink J, Konigsrainer A, Mohammad O, Jakobs R, Willis S, Demir IE, Friess H, Hetjens S, Ebert MP, Reissfelder C, Vassilev G. Conservative versus surgical therapy for idiopathic and secondary megacolon or megarectum in adults - a retrospective multicentre controlled study. Z Gastroenterol. 2024 Nov;62(11):1913-1923. doi: 10.1055/a-2360-5008. Epub 2024 Sep 11. PMID 39260392